CLINICAL TRIAL: NCT03165344
Title: Effectiveness Evaluation of Mixed Gel of Hydrocortisone and Aluminium Phosphate Preventing Endoscopic Submucosal Dissection Postoperative Stenosis for Patients With Early Esophageal Cancer Invading More Than 2/3 Esophageal Perimeter
Brief Title: Mixed Gel of Hydrocortisone and Aluminium Phosphate Preventing Endoscopic Submucosal Dissection Postoperative Stenosis for Patients With Large Esophageal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Huang Yonghui, Chief physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Z171100001017091
Record Dates: First submitted 2017-04-07; First posted 2017-05-24 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Esophageal Stenosis Acquired
MeSH Terms: interventions — Drug Administration Routes; Triamcinolone Acetonide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrocortisone group (Experimental)
  Interventions: Other: Hydrocortisone sodium succinate mixed with Aluminium Phosphate gel (route of administration)
- prednisone grope (Placebo Comparator)
  Interventions: Other: Triamcinolone Acetonide (route of administration); Other: Prednisone (route of administration)

INTERVENTIONS:
Other: Hydrocortisone sodium succinate mixed with Aluminium Phosphate gel (route of administration) — the test group begin to take hydrocortisone sodium succinate mixed with Aluminium Phosphate gel after 24 hours and gradually reduse the dose.
  Arms: hydrocortisone group
Other: Triamcinolone Acetonide (route of administration) — The control group will get local injection of triamcinolone acetonide in wound during the operation.
  Arms: prednisone grope
Other: Prednisone (route of administration) — The control group begin to take oral prednisone after 24 hours and gradually reduse the dose.
  Arms: prednisone grope

SUMMARY:
Endoscopic submucosal dissection as the fastest growing endoscopic treatment technology in the past decade has been widely used in the treatment of early esophageal cancer and gastric cancer without local lymph node metastasis. The main complications of ESD treatment of early esophageal cancer are hemorrhage, perforation, postoperative esophageal stenosis, infection, etc. Postoperative esophageal stenosis is the most common and major complication after ESD treating patients with lesion involving more than 2/3 esophagus cycle. It is very important to prevent esophageal stricture after ESD. Glucocorticoid is gradually concerned by clinical research because it can inhibit local inflammatory response and reduce the formation of connective tissue in order to prevent postoperative stenosis. The specific usages include endoscopic injection of corticosteroids, oral corticosteroids and combination of them. The study shows that the incidence of esophageal stricture after using glucocorticoid can be reduced effectively. Currently, there is no uniform consensus on the use of glucocorticoids, such as specific drugs, dosage, course of treatment, route of administration. In particular, efficacy comparison of different routes of administration is laking. Studies have shown that endoscopic injection triamcinolone acetonide in some patients with intractable esophageal stricture is not very effective, but it can be treated with oral corticosteroids. Aluminium Phosphate Gel is a kind of neutral buffer. The main component aluminum phosphate can form a strong ion buffer system in acidic environment. The structure of its auxiliary components agar and pectin is similar to that of natural mucus. It forms a mucous layer in the esophagus to restore and protect the esophageal mucosa. Therefore, investigators assume the hydrocortisone sodium succinate aluminum phosphate mixed gel can be used for preventing postoperative ESD stenosis of patients with a large area of early esophageal cancer. This study will design a randomized controlled trial to compare the effect of oral hydrocortisone sodium succinate mixed Aluminium Phosphate Gel and local injection of triamcinolone acetonide plus oral prednisone for the prevention of ESD postoperative esophageal stricture in patients with a large area of early esophageal cancer.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection as the fastest growing endoscopic treatment technology in the past decade has been widely used in the treatment of early esophageal cancer and gastric cancer without local lymph node metastasis. The main complications of ESD treatment of early esophageal cancer are hemorrhage, perforation, postoperative esophageal stenosis, infection, etc. Postoperative esophageal stenosis is the most common and major complication after ESD treating patients with lesion involving more than 2/3 esophagus cycle. It is very important to prevent esophageal stricture after ESD. Glucocorticoid is gradually concerned by clinical research because it can inhibit local inflammatory response and reduce the formation of connective tissue in order to prevent postoperative stenosis. The specific usages include endoscopic injection of corticosteroids, oral corticosteroids and combination of them. The study shows that the incidence of esophageal stricture after using glucocorticoid can be reduced effectively. Currently, there is no uniform consensus on the use of glucocorticoids, such as specific drugs, dosage, course of treatment, route of administration. In particular, efficacy comparison of different routes of administration is laking. Studies have shown that endoscopic injection triamcinolone acetonide in some patients with intractable esophageal stricture is not very effective, but it can be treated with oral corticosteroids. Aluminium Phosphate Gel is a kind of neutral buffer. The main component aluminum phosphate can form a strong ion buffer system in acidic environment. The structure of its auxiliary components agar and pectin is similar to that of natural mucus. It forms a mucous layer in the esophagus to restore and protect the esophageal mucosa. Therefore, investigators assume the hydrocortisone sodium succinate aluminum phosphate mixed gel can be used for preventing postoperative ESD stenosis of patients with a large area of early esophageal cancer. This study will design a randomized controlled trial to compare the effect of oral hydrocortisone sodium succinate mixed Aluminium Phosphate Gel and local injection of triamcinolone acetonide plus oral prednisone for the prevention of ESD postoperative esophageal stricture in patients with a large area of early esophageal cancer.

The investigators will recruit patients according to admission criteria and exclusion criteria. The patients will be randomly divided into oral hydrocortisone mixed Aluminium Phosphate gel group (experimental group) and local injection of triamcinolone acetonide plus oral prednisone group (control group). The test group begin to take hydrocortisone sodium succinate mixed with Aluminium Phosphate gel after 24 hours and gradually reduse the dose. The control group will get local injection of triamcinolone acetonide in wound during the operation, and begin to take oral prednisone after 24 hours and gradually reduse the dose. The main result is esophageal stenosis rate 3 months after ESD.

ELIGIBILITY:
Inclusion Criteria:

1. early esophagus cancer,lesions confined to the mucosal layer,ESD treatment is feasible and the resection range is ≥ 2/3 esophageal perimeter
2. age 18 years or older
3. chest CT scan without lymph node metastasis

Exclusion Criteria:

1. patients with early esophagus cancer do not agree with endoscopic treatment
2. occurrence of perforation in ESD requires further treatment
3. lesions invading the muscularis mucosa and below
4. postoperative pathologic assessment of ESD prompting incomplete resection and requiring radiotherapy and chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Esophageal stenosis rate | 3 months after ESD
  Esophageal stenosis is defined as that the standard upper gastrointestinal endoscopy with the diameter of 9.2mm can not pass the esophageal lumen.

SECONDARY OUTCOMES:
The rate of endoscopic balloon dilation and its therapeutic effect. | 3 months after ESD
  We will compare the rate of endoscopic balloon dilation and its therapeutic effect of the two groups
Healing condition of the wound | 3 months after ESD
  healing rate=（area of wound after surgery - remained wound area）/area of wound after surgery
Side effect of drugs | 3 months after ESD
  including hypertension、hyperglycemia、electrolyte imbalance etc

CONTACTS AND LOCATIONS:
Overall Officials: Yonghui Huang, archiater, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Result] Merkow RP, Bilimoria KY, Keswani RN, Chung J, Sherman KL, Knab LM, Posner MC, Bentrem DJ. Treatment trends, risk of lymph node metastasis, and outcomes for localized esophageal cancer. J Natl Cancer Inst. 2014 Jul 16;106(7):dju133. doi: 10.1093/jnci/dju133. Print 2014 Jul. PMID 25031273
- [Result] Mizuta H, Nishimori I, Kuratani Y, Higashidani Y, Kohsaki T, Onishi S. Predictive factors for esophageal stenosis after endoscopic submucosal dissection for superficial esophageal cancer. Dis Esophagus. 2009;22(7):626-31. doi: 10.1111/j.1442-2050.2009.00954.x. Epub 2009 Mar 6. PMID 19302207
- [Result] Ono S, Fujishiro M, Niimi K, Goto O, Kodashima S, Yamamichi N, Omata M. Predictors of postoperative stricture after esophageal endoscopic submucosal dissection for superficial squamous cell neoplasms. Endoscopy. 2009 Aug;41(8):661-5. doi: 10.1055/s-0029-1214867. Epub 2009 Jun 29. PMID 19565442
- [Result] Shi Q, Ju H, Yao LQ, Zhou PH, Xu MD, Chen T, Zhou JM, Chen TY, Zhong YS. Risk factors for postoperative stricture after endoscopic submucosal dissection for superficial esophageal carcinoma. Endoscopy. 2014 Aug;46(8):640-4. doi: 10.1055/s-0034-1365648. Epub 2014 May 15. PMID 24830402
- [Result] Hochberger J, Koehler P, Wedi E, Gluer S, Rothstein RI, Niemann H, Hilfiker A, Gonzalez S, Kruse E. Transplantation of mucosa from stomach to esophagus to prevent stricture after circumferential endoscopic submucosal dissection of early squamous cell. Gastroenterology. 2014 Apr;146(4):906-9. doi: 10.1053/j.gastro.2014.01.063. Epub 2014 Feb 8. No abstract available. PMID 24512802
- [Result] Machida H, Tominaga K, Minamino H, Sugimori S, Okazaki H, Yamagami H, Tanigawa T, Watanabe K, Watanabe T, Fujiwara Y, Arakawa T. Locoregional mitomycin C injection for esophageal stricture after endoscopic submucosal dissection. Endoscopy. 2012 Jun;44(6):622-5. doi: 10.1055/s-0032-1306775. Epub 2012 May 25. PMID 22638783
- [Result] Yamaguchi N, Isomoto H, Nakayama T, Hayashi T, Nishiyama H, Ohnita K, Takeshima F, Shikuwa S, Kohno S, Nakao K. Usefulness of oral prednisolone in the treatment of esophageal stricture after endoscopic submucosal dissection for superficial esophageal squamous cell carcinoma. Gastrointest Endosc. 2011 Jun;73(6):1115-21. doi: 10.1016/j.gie.2011.02.005. Epub 2011 Apr 14. PMID 21492854
- [Result] Hanaoka N, Ishihara R, Takeuchi Y, Uedo N, Higashino K, Ohta T, Kanzaki H, Hanafusa M, Nagai K, Matsui F, Iishi H, Tatsuta M, Ito Y. Intralesional steroid injection to prevent stricture after endoscopic submucosal dissection for esophageal cancer: a controlled prospective study. Endoscopy. 2012 Nov;44(11):1007-11. doi: 10.1055/s-0032-1310107. Epub 2012 Aug 28. PMID 22930171
- [Result] Hashimoto S, Kobayashi M, Takeuchi M, Sato Y, Narisawa R, Aoyagi Y. The efficacy of endoscopic triamcinolone injection for the prevention of esophageal stricture after endoscopic submucosal dissection. Gastrointest Endosc. 2011 Dec;74(6):1389-93. doi: 10.1016/j.gie.2011.07.070. PMID 22136782
- [Result] Morikawa N, Honna T, Kuroda T, Watanabe K, Tanaka H, Takayasu H, Fujino A, Tanemura H, Matsukubo M. High dose intravenous methylprednisolone resolves esophageal stricture resistant to balloon dilatation with intralesional injection of dexamethasone. Pediatr Surg Int. 2008 Oct;24(10):1161-4. doi: 10.1007/s00383-008-2224-7. PMID 18704454
- [Result] Hishiki T, Kouchi K, Saito T, Terui K, Sato Y, Mitsunaga T, Nakata M, Yoshida H. Successful treatment of severe refractory anastomotic stricture in an infant after esophageal atresia repair by endoscopic balloon dilation combined with systemic administration of dexamethasone. Pediatr Surg Int. 2009 Jun;25(6):531-3. doi: 10.1007/s00383-009-2367-1. Epub 2009 May 9. PMID 19430800